CLINICAL TRIAL: NCT00671866
Title: Neurotoxic Health Hazards of Long-Term Low-Level Exposure to Organophosphate (OP) Compounds in in Hula Valley
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: y.finkelstein.ctil.
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2008-04

CONDITIONS: Peripheral Neuropathy
Keywords: OP; Pesticides; Long-Term Low Level Exposure; Occupational Health; Neurobehavioral Effects
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- 1: Agricultural Workers
- 2: Non - Agricultural Workers
- 3: Kibbitz Residents working else where

SUMMARY:
During 1987-1991, WHO supported studies of exposures and short term neurobehavioral effects in a cohort (n=200) with occupational and community exposures to pesticide drift containing organophosphates from orchards and cotton fields in the Hula Valley. We aim (1) to re-examine neurobehavioral outcomes in members of the original cohort and (2) to examine cognitive effects in children with residential exposures. In adults, we will carry out assays of alkyl phosphates, PON1 (paraoxonase-1), NTE (Neuropathy Target Esterase), neurobehavioral tests of cognitive and performance skills, nerve conduction measurements and mood status. We will carry out Psycho-Didactic tests in children. The findings will advance knowledge on delayed term health effects of lengthy everyday exposure to OP pesticides and guide regulatory policy.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the former study twenty years ago

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Kibbutzim
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology and Toxicology Unit and Service, Shaare Zedek Med Ctr, Jerusalem, Israel